CLINICAL TRIAL: NCT06884969
Title: Investigation of Motor Development and Sensory Processing Skills in Infants With a History of Late-onset Sepsis
Brief Title: Late-onset Sepsis and Development
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Nigde Omer Halisdemir University
Other Study IDs: late-onset sepsis
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-03

CONDITIONS: Sepsis Newborn; Motor Development; Sensory Integration Dysfunction
Keywords: sepsis; motor development; sensory processing skills; infant
MeSH Terms: conditions — Neonatal Sepsis; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Late-onset sepsis: Neonatal sepsis is a common condition that triggers both pro- and anti-inflammatory responses in the organism, affects various tissues, and alters enzymatic activities. Immaturity of the immune system, the use of central catheters during parenteral nutrition, and delayed enteral feeding with breast milk are known risk factors for late-onset sepsis in neonates. Late-onset sepsis is defined as sepsis that occurs after the first 72 hours of postnatal life and is characterized by the presence of infectious symptoms (such as fever, irritability, lethargy, apnea, growth retardation, feeding refusal, tachycardia, or tachypnea), acute-phase reactants (elevated interleukin-6 or C-reactive protein), and/or a positive blood culture accompanied by leukopenia.
  The planned study will include toddlers with a history of late-onset sepsis, focusing on the 10-18 month period.
  Interventions: Behavioral: Test of Sensory Function in Infants; Behavioral: Peabody Motor Development Scale-2
- Healthy infants: A control group consisting of healthy babies, born at term and between 10-18 months of age, with no history of sepsis will be created.
  Interventions: Behavioral: Test of Sensory Function in Infants; Behavioral: Peabody Motor Development Scale-2

INTERVENTIONS:
Behavioral: Test of Sensory Function in Infants — It was planned to use the Test of Sensory Function in Infants to evaluate the sensory development of infants. Test of sensory function in infants is frequently used to evaluate the sensory processing functions of infants aged 4-18 months.
Behavioral: Peabody Motor Development Scale-2 — Peabody Motor Development Scale-2 was planned to be used to assess motor development. Peabody Motor Development Scale-2 was designed to determine developmental delays in children between 0-72 months.

SUMMARY:
Neonatal sepsis is classified as early-onset and late-onset sepsis. Early-onset sepsis occurs within the first 72 hours after birth and is associated with a mortality rate of 10-15%. Late-onset sepsis, on the other hand, is characterized by its onset after the first 72 hours of life in infants who have been exposed to microorganisms in the postnatal environment. Preterm infants are the most vulnerable group in terms of sepsis, and the incidence of hospital-acquired late-onset sepsis can reach up to 40% in extremely preterm neonates. In contrast, community-acquired late-onset sepsis has been predominantly reported in late preterm and full-term infants. Community-acquired late-onset sepsis is the most common form of sepsis among term neonates and accounts for half of all sepsis episodes in infants born at ≥37 weeks of gestation.During infancy, particularly when children begin to crawl and walk, they actively explore their environment and attempt to expand their motor repertoire. However, when examining studies related to sepsis, it appears that assessments conducted during the walking infant period are quite limited, with most research focusing on school-aged and preschool children. Furthermore, existing studies primarily address behavioral problems and motor performance issues.Therefore, considering that this period represents an early stage of development, it is planned to include infants aged 10 to 18 months in the present study. The aim of this study is to evaluate the motor development and sensory processing skills of infants with a history of sepsis and to compare them with their healthy peers without a history of sepsis.

DETAILED DESCRIPTION:
Neonatal sepsis is a common condition that triggers both pro- and anti-inflammatory responses in the organism, affects various tissues, and alters enzymatic activities. Immaturity of the immune system, the use of central catheters during parenteral nutrition, and delayed enteral feeding with breast milk are well-known risk factors for late-onset sepsis in neonates. Late-onset sepsis is defined as sepsis that occurs after 72 hours of postnatal life and is characterized by infectious symptoms (such as fever, irritability, lethargy, apnea, growth retardation, feeding refusal, tachycardia, or tachypnea), the presence of acute phase reactants (elevated interleukin-6 or C-reactive protein), and/or positive blood culture and leukopenia criteria. The evaluation of sensory processing skills becomes crucial in children aged 10 to 18 months, a period when they begin to explore their environment through walking and trial-and-error learning. Motor development during this period largely depends on active trial-and-error learning, making effective sensory processing a critical component. However, the first two years of life, which represent the fastest and most critical period of development, have been largely neglected in terms of assessing motor and sensory processing abilities in these children.The planned study aims to address this gap by focusing on the 10- to 18-month period, evaluating motor development and sensory processing skills in infants with a history of sepsis during the early walking stage. This unique approach may provide valuable insights into the early diagnosis and intervention processes for developmental problems.

ELIGIBILITY:
Inclusion Criteria:

* Term infants with a history of late-onset sepsis
* Post-term infants between 10-18 months

Exclusion Criteria:

* History of early neonatal sepsis,
* Preterm infants,
* Those with congenital infection or proven genetic alterations,
* Infants diagnosed with metabolic, neurological and genetic diseases,
* Children whose parents do not volunteer for the study

Ages: 10 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Late-onset sepsis is defined as sepsis that occurs after 72 hours of postnatal life and meets criteria for infectious symptoms and the presence of acute-phase reactants and/or leukopenia with positive blood cultures. The planned study aims to address the lack of evaluation of motor development and sensory processing skills in toddlers with a history of sepsis by focusing on the 10-18 month period. This unique approach may shed light on the early diagnosis and intervention processes of developmental problems.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales | Second Edition (PDMS-2) | 10-18 months
  Peabody Motor Development Scale-2 was planned to be used to evaluate motor development. Peabody Motor Development Scale-2 was designed to determine developmental delays in children between 0-72 months. Separate tests and rating scales for both gross motor skills and fine motor skills were used to evaluate children's motor development.
Test of Sensory Functions in Infants | 10-18 months
  It was planned to use the Test of Sensory Function in Infants. The Test of Sensory Function in Infants is frequently used to evaluate the sensory processing functions of infants aged 4-18 months. It is used to determine whether an infant has a sensory processing problem and to what extent. It consists of 24 items. The Test of Sensory Function in Infants requires the infant to be stimulated and interacted with various materials. The total score varies between 0-49 and the test has normative values for different age groups. Although it is used from the fourth month onwards, the most reliable and valid results are obtained between 7-18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia ZORLULAR, Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folio, M.R., Peabody developmental motor scales. DLM Teaching Resources, 1983.
- [Background] DeGangi, G.A. and S.I. Greenspan, The development of sensory functions in infants. Physical & Occupational Therapy in Pediatrics, 1989. 8(4): p. 21-33.
- [Background] Stoll BJ, Hansen NI, Adams-Chapman I, Fanaroff AA, Hintz SR, Vohr B, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental and growth impairment among extremely low-birth-weight infants with neonatal infection. JAMA. 2004 Nov 17;292(19):2357-65. doi: 10.1001/jama.292.19.2357. PMID 15547163
- [Background] Greenhow TL, Hung YY, Herz AM. Changing epidemiology of bacteremia in infants aged 1 week to 3 months. Pediatrics. 2012 Mar;129(3):e590-6. doi: 10.1542/peds.2011-1546. Epub 2012 Feb 27. PMID 22371459
- [Derived] Zorlular R, Degirmencioglu H, Zorlular A. Sensory processing and motor development in term infants following late-onset neonatal sepsis-a cross-sectional study. Eur J Pediatr. 2025 Nov 1;184(11):726. doi: 10.1007/s00431-025-06571-1. PMID 41175143